CLINICAL TRIAL: NCT03832803
Title: Less to Hold - A Comparison of Bladder Toxicities (Side Effects) in Patients Undergoing Prostate Radiotherapy Between Patients Treated With Empty Bladder and Those on a Drinking Protocol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2113
Record Dates: First submitted 2019-01-29; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: 50 patients receiving radical radiotherapy to the prostate were randomised using 1:1 into 2 groups. Group A followed the conventional drinking protocol at our centre (200ml prior to treatment) and group B were treated with an empty bladder. Baseline, end of treatment and 6 week follow up scores were prospectively collected for IPSS, LENT SOMA bowel toxicity and quality of life questionnaires.
Masking Description: Investigator masking for randomisation purposes only. Masking not possible for intervention whilst on treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empty Bladder (Experimental): Empty bladder prior to treatment.
  Interventions: Behavioral: Empty bladder
- Full Bladder (Other): Conventional drinking protocol - 200ml water prior to treatment.
  Interventions: Behavioral: Full bladder

INTERVENTIONS:
Behavioral: Empty bladder — No drinking protocol.
  Arms: Empty Bladder
Behavioral: Full bladder — Followed drinking protocol
  Arms: Full Bladder

SUMMARY:
Radical radiotherapy to the prostate is conventionally treated with a full bladder with the aim of minimising dose to the bladder and small bowel to prevent significant side effects. Tolerance of the bladder filling protocol varies depending on patients' baseline urinary function. It is not uncommon for some men to have "accidents" during treatment causing understandable distress. This can also extend the treatment time and cause knock on delays in the radiotherapy department.

Several United Kingdom (UK) centres report treating with an empty bladder. The investigators carried out a feasibility study comparing treatment with full bladder to empty bladder to ascertain if the investigators can safely change our protocol to that of an empty bladder.

DETAILED DESCRIPTION:
50 patients receiving radical radiotherapy to the prostate were randomised using closed envelope technique 1:1 into 2 groups. Group A followed the conventional drinking protocol at our centre (200ml prior to treatment) and group B were treated with an empty bladder. Baseline, end of treatment and 6 week follow up scores were prospectively collected for International prostate Symptom Score(IPSS), Late Effects Normal Tissue Task Force - Subjective, Objective, Management, Analytic (LENT SOMA) bowel toxicity and quality of life questionnaires. The investigators also looked at bowel and bladder Dose Volume Histogram (DVH) to ensure constraints were met.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer receiving radical radiotherapy.

Exclusion Criteria:

* Not nodal disease.
* Not prostate bed radiotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Change in IPSS score | Baseline to end of treatment (4 weeks or 7 and a half weeks depending on radiotherapy schedule); to 6 week follow up; and to 1 year follow up.
  IPSS - The International Prostate Symptom Score is a 7 question scale which assesses urinary toxicity. Each question is scored 0-5 totalling a maximum score of 35. A score of 0-7 correlates to mildly symptomatic; 8-19, moderately symptomatic; 20-35, severely symptomatic.

SECONDARY OUTCOMES:
Change in LENT SOMA score | Baseline to end of treatment (4 weeks or 7 and a half weeks depending on radiotherapy schedule); to 6 week follow up; and to 1 year follow up.
  LENT SOMA - The Late Effects in Normal Tissues Subjective, Objective, Management and Analytic Scales. This is a questionnaire that assesses individual bowel symptoms asking initially whether or not they occur and then scoring the frequency, the higher the score, the more frequent the event. Each question has it's own range of score which is explained on the questionnaire. The scores will be compared for individual questions and there will not be any combining of scores between questions.
Bowel and bladder DVH | At time of radiotherapy planning scan which happens at baseline, on day of randomisation.
  Dose to bowel and bladder is calculated and documented if it meets the optimal or mandatory constraints

CONTACTS AND LOCATIONS:
Overall Officials: Alison Birtle, Principal Investigator — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (1):
- Lancashire Teaching Hospitals NHS Foundation Trust, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No